CLINICAL TRIAL: NCT03414463
Title: Training to Reconnect With Emotional Awareness Therapy
Acronym: TREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Flora Hammond, Chair of Department of Physical Medicine and Rehabilitation, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1711946589
Record Dates: First submitted 2018-01-11; First posted 2018-01-30 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury; Alexithymia
Keywords: Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Affective Symptoms; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREAT (Experimental): A 4-week one-to-one intervention between the clinical RA (cRA) and participant. Comprised of eight sessions, it involves psycho-educational lessons and skill-building exercises to achieve objectives based on the characteristics of alexithymia.
  Interventions: Behavioral: TREAT
- Waitlist Control (Experimental): After Time 1 testing in Week 1, participants randomized to WLC will not receive any treatment during Weeks 2-5. The only staff interaction during this no treatment time period will be to schedule Time 2 testing appointment for week 6. After Time 2 testing, WLC will receive TREAT (weeks 14-17), followed up with testing.
  Interventions: Behavioral: TREAT

INTERVENTIONS:
Behavioral: TREAT — A 4-week one-to-one intervention between the clinical RA (cRA) and participant. Comprised of eight sessions, it involves psycho-educational lessons and skill-building exercises to achieve objectives based on the characteristics of alexithymia.

SUMMARY:
To decrease emotional self-awareness deficits and improve emotional self-regulation, particularly anxiety, anger, depression, and positive affect, through the treatment of alexithymia.

DETAILED DESCRIPTION:
Phase II randomized, Waitlist Control (WLC) trial with 3-month follow-up to further establish proof of concept and early efficacy of TREAT (1:1 alexithymia treatment) for post-TBI alexithymia. It is anticipated that our target sample size is 44. The purpose of this study is to examine differences in post-treatment self-reported alexithymia and emotional self-awareness in participants with TBI randomized to TREAT or WLC. In addition to examining the differences in post-treatment self-reported emotion regulation (general), anxiety, anger, depression, positive affect (PA), global emotional function and quality of life in participants with TBI randomized to TREAT or WLC.

ELIGIBILITY:
Inclusion Criteria:

* TBI (injury due to a external physical force)
* Complicated mild, moderate, or severe TBI (defined by Glasgow Coma Scale (GCS) in Emergency Department (ED) (≤12), or Post traumatic amnesia (PTA) (≥1 day),Loss of Conscientious (LOC) (≥30 minutes),or positive head CT scan consistent with TBI)
* At least 18 years or older
* ≥1 year post-injury
* Adequate vision, hearing, speech, and comprehension
* Reliable mode of transportation
* Available for treatment during regular business hours
* Have moderate to high screening alexithymia score (TAS-20 ≥52)
* If participating in active psychological treatment prior to enrollment, their participation must be ongoing for 4 or more weeks

Exclusion Criteria:

* Diagnosed with pre-morbid neurological disorder that could affect mood and cognition (e.g., stroke, Alzheimer's disease, Parkinson's disease); does not include controlled seizures
* Diagnosed with major psychiatric disorder (e.g., schizophrenia, Borderline Personality Disorder)
* Severe Depression and/or perceived risk to self or others
* Developmental disability (e.g. autism, developmental delay)
* Unstable or anticipated medication changes related to mood or emotion during study participation
* Having started psychological treatment less than 4 weeks prior to enrollment
* Actively participating in the Traumatic Brain Injury Model System (TBIMS) alexithymia outcome module

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Change in Toronto Alexithymia Scale-20 (TAS-20) | Baseline Week , 6, 18, 30
  This is a 20-item self report questionnaire comprised of three sub-constructs (Difficulty Identifying feelings, Difficulty Describing feelings, Externally-oriented Thinking). The full scale range is 20-100 (higher scores indicate higher alexithymia). Subscales are summed to compute a total score. Scores between 52 and 60 indicate moderate alexithymia; scores 61 and higher indicate high alexithymia.
Change in Levels of Emotional Awareness Scale (LEAS) | Baseline Week , 6, 18, 30
  objective, performance-based measure of emotional awareness and labeling. Short hypothetical scenarios are presented and participants are asked to describe how they and others would feel in the context of the scenarios. Participants' responses are scored with an electronic system, removing human bias and interpretation. The LEAS has parallel forms (A and B), which will alternate at testing sessions.

SECONDARY OUTCOMES:
Difficulty with Emotion Regulation Scale (DERS) | Baseline Week , 6, 18, 30
  Using a 5-point Likert scale, participants rate the frequency they utilize self-regulation behaviors in response to general emotional distress. There are 6 subscales: Lack of Emotional Awareness, Lack of Emotional Clarity, Difficulties Controlling Impulsive Behaviors When Distressed, Difficulties Engaging in Goal-Directed Behavior When Distressed, Non-acceptance of Negative Emotional Responses, and Limited Access to Effective Emotion Regulation Strategies. Items are summed to provide a Total Emotion Dysregulation score. The DERS has high internal consistency, test-retest reliability, and good construct validity.61 Importantly, because this measure assesses difficulties regulating all types of emotions, it captures different information than that provided by measures specific to anxiety, anger, or depression which can miss more general, yet common, self-regulation problems.
Generalized Anxiety Disorder Assessment (GAD-7): | Baseline Week , 6, 18, 30
  A self-report 7-item questionnaire (score range is 0 to 21) that assesses frequency of seven anxiety symptoms linked to the DSM-IV criteria for Generalized Anxiety Disorder (GAD). Higher scores indicate higher levels of anxiety severity (higher=worse).
Patient Health Questionnaire 9 (PHQ-9) | Baseline Week , 6, 18, 30
  This self-report depression assessment uses a 3-point Likert scale (maximum score 27), with established validity and reliability, including in the TBI population. Participants rate the frequency of specified problems during the past 2 weeks.
State-Trait Anger Expression Inventory (STAXI) | Baseline Week , 6, 18, 30
  consists of 57 questions that address the intensity and the frequency of internal and external expressions of anger rated on a 4-point Likert scale. The measure is comprised of 3 subscales, each with individual t-scores: "How I feel right now"; "How I generally feel"; "How I generally react or behave when angry or furious." For the purpose of this study, we will only be administering the latter 2 subscales ("How I generally feel" and "How I generally react or behave).
Positive and Negative Affect Scale (PANAS) | Baseline Week , 6, 18, 30
  20-item subjective assessment of mood (10 items for Positive Affect and 10 for Negative Affect). Participants rate on a 5-point scale the extent to which they have experienced each mood state during a specified time frame. This measure showed a significantly increased positive affect in Phase I. The measure has shown good test-retest reliability over a number of weeks and validity in a variety of populations
Patient Global Impression of Change (PGIC) | Week 6 or 18 depending on randomization
  This Likert scale, used in prior TBI studies captures the patient perspectives of clinically important change in participant global emotional function and quality of life during the course of study participation. Responses range from 1 (very much worse) to 7 (very much improved). Depending on participants' preferences
Caregiver Global Impression of Change (CaGIC) | Week 6, 18, 30
  This Likert scale, used in prior TBI studies captures the caregiver perspectives of clinically important change in participant global emotional function and quality of life during the course of study participation. Responses range from 1 (very much worse) to 7 (very much improved). Depending on participants' preferences
Participant Satisfaction | Week 6 or 18 depending on randomization
  Using the same satisfaction questions from the Phase I preliminary study, participants will respond to the following statements using a 5-point Likert scale (1=Strongly Disagree to 5=Strongly Agree): 1) I am satisfied with the information taught in this training program; 2) The lessons taught in the training are relevant to my needs; 3) I will try to use the lessons I learned from this training in my daily life; 4) The information provided in this training program was easy to understand; 5) If a friend or family member was in need similar help, I would recommend the program to him or her; and 6) I think the training program helped me to deal more effectively with my emotions. The participant will be asked seventh open-ended questions regarding additional comments about the training program. Depending on participants' preferences

CONTACTS AND LOCATIONS:
Overall Officials: Flora Hammond, MD, Principal Investigator — Indiana University
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States